CLINICAL TRIAL: NCT06372080
Title: The Effects of Resistance Training With Hydrolyzed Collagen Supplementation on Muscle and Tendon Adaptation in Healthy Young Adults
Brief Title: Resistance Training and Hydrolyzed Collagen Supplementation in Healthy Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 19/SPS/054
Record Dates: First submitted 2024-04-03; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-02

CONDITIONS: Healthy Participants; Nutrition; Exercise Training
Keywords: hydrolyzed collagen; tendon properties; maximal strength; muscle size; resistance exercise
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: The study design is a single-blind (participants were unaware of their group allocation), randomized controlled trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance training with hydrolyzed collagen ingestion in healthy young men (Experimental): Healthy young men, pair-matched by age, body mass, height, and baseline strength, will be randomly allocated to the collagen (COL) or placebo (PLA) group.
  Pre- and post-training assessments are patellar tendon properties, maximal knee flexor and extensor strengths and vastus lateralis muscle morphology using an isokinetic dynamometer and ultrasound scan.
  Participants will perform the 10-week progressive resistance training program three times per week and training loads will be adjusted weekly based on the prior session's performance.
  In each session, two different calorie-matched beverages were given immediately before the start of resistance training. 30 grams of hydrolyzed collagen (HC) and 30.5 grams of maltodextrin were used for COL and PLA respectively. HC or maltodextrin was mixed with 250 milliliters of water, 50 milligrams of vitamin C and 3 grams non-caloric sweetener which was used to mask flavour in an opaque bottle.
  Interventions: Dietary Supplement: Resistance training with hydrolyzed collagen ingestion in healthy young men
- Resistance training with hydrolyzed collagen ingestion in healthy young women (Experimental): The intervention procedure is the same as for Arm 1 except that the participants will be healthy young women (not men).
  Interventions: Dietary Supplement: Resistance training with hydrolyzed collagen ingestion in healthy young women

INTERVENTIONS:
Dietary Supplement: Resistance training with hydrolyzed collagen ingestion in healthy young men — Participants in this intervention will be healthy young men. The information of nutritional supplements is below.
  Hydrolyzed collagen: 30 grams unflavored hydrolysed collagen (HC) (Myprotein, Cheshire, UK) 30.5 grams unflavored maltodextrin (Myprotein, Cheshire, UK) 50 milligrams vitamin C powder (Holland and Barrett Retail Limited, Warwickshire, UK) 3 grams non-caloric sweetener (Truvia®, SilverSpoon, London, UK)
  Arms: Resistance training with hydrolyzed collagen ingestion in healthy young men
Dietary Supplement: Resistance training with hydrolyzed collagen ingestion in healthy young women — Participants in this intervention will be healthy young women. The same nutritional supplements in Arm 1 wil be used in Arm 2.
  Arms: Resistance training with hydrolyzed collagen ingestion in healthy young women

SUMMARY:
The goal of this clinical trial is to investigate the effects of resistance training with hydrolyzed collagen ingestion on changes in muscle and tendon adaptation in healthy young men and women.

The main questions it aims to answer are:

* Does resistance training with hydrolyzed collagen ingestion lead to greater changes in tendon properties than resistance training alone?
* Does resistance training with hydrolyzed collagen ingestion lead to greater changes in muscle size than resistance training alone?

Participants will be randomly assigned to collagen or placebo groups. Participants will perform resistance training three times per week for 10 weeks and hydrolyzed collagen or maltodextrin will be given to collagen or placebo group respectively immediately before each resistance training session. Also, vitamin C will be given to both groups.

Researchers will compare collagen and placebo groups to see if hydrolyzed collagen ingestion with resistance exercise would have beneficial effects on changes in muscle and tendon more than resistance training alone. Therefore, using isokinetic dynamometer and ultrasonography, maximal leg strength, morphological, mechanical, and material properties of the patellar tendon and vastus lateralis muscle size and architecture will be assessed.

DETAILED DESCRIPTION:
Young, healthy, active men and women will ingest 30 grams of hydrolyzed collagen or a calorie matched beverage (maltodextrin) alongside vitamin C prior to performing high-intensity resistance training 2 - 3 times per week for 10 weeks.

The aim of this study is to investigate the effect of combining hydrolyzed collagen supplementation with resistance training in young men and women. If supplementation with hydrolyzed collagen leads to a greater change in tendon size, stiffness, and Young's modulus than resistance training alone, this will allow us to recommend this type of intervention to young athletes seeking to improve tendon health and/or athletic performance.

The experimental design and measurements will be the same in the Arm 1 and Arm 2 but the differences will be sex where participants in Arm 1 will be healthy young men while participants in Arm 2 will be healthy young women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young male or female
* No history of patellar tendon injuries in the past 6 months
* No history of lower limb musculoskeletal injuries in the past 6 months
* Non-smokers (including e-cigarettes)
* Free from cardiovascular and metabolic diseases
* Nullipara (a woman who has never given birth)

Exclusion Criteria:

* Age less than 18 years or higher than 40 years
* Being vegan or vegetarian (due to the mammalian source of collagen)
* Consumption of nutritional supplementation that purportedly affects muscle-tendon adaptation or recovery (i.e. protein powder, vitamin C, collagen)
* BMI over 30 kg/m2
* Previous anterior cruciate ligament injury where the patellar tendon was used as a graft

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Maximal knee extensor (quadriceps) muscle strength | 12 weeks (10 weeks' intervention plus one week either side for assessments)
  Using isokinetic dynamometer, knee extensor maximal isometric voluntary contraction torque (in Newton meters) will be measured.
Maximal knee flexor (hamstring) muscle strength | 12 weeks (10 weeks' intervention plus one week either side for pre- and post-intervention assessments)
  Using an isokinetic dynamometer, knee flexor maximal isometric voluntary contraction torque (in Newton meters) will be measured.
Patellar tendon cross-sectional area | 12 weeks (10 weeks' intervention plus one week either side for pre- and post-intervention assessments)
  Using ultrasonography, patellar tendon cross-sectional area (in millimeters squared) will be measured.
Patellar tendon stiffness | 12 weeks (10 weeks' intervention plus one week either side for pre- and post-intervention assessments)
  Using ultrasonography, patellar tendon stiffness (in Newtons per millimeter) will be measured.
Vastus lateralis (VL) muscle size | 12 weeks (10 weeks' intervention plus one week either side for pre- and post-intervention assessments)
  Using ultrasonography, the VL anatomical cross-sectional area (in centimeters squared) will be measured.
Vastus lateralis (VL) muscle fascicle length | 12 weeks (10 weeks' intervention plus one week either side for pre- and post-intervention assessments)
  Using ultrasonography, VL muscle fascicle length (in millimeters) will be measured.
Vastus lateralis (VL) muscle fascicle pennation angle | 12 weeks (10 weeks' intervention plus one week either side for pre- and post-intervention assessments)
  Using ultrasonography, VL muscle fascicle pennation angle (in degrees) will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute for Sport and Exercise Sciences, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No